CLINICAL TRIAL: NCT05106036
Title: Preventing Cognitive Decline by Reducing BP Target Trial
Acronym: PCOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Duke University (Other); Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Miguel Vazquez, Professor, Clinical Director, Division of Nephrology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU-2021-0735; R33AG068486 (NIH)
Record Dates: First submitted 2021-09-27; First posted 2021-11-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Decline; Blood Pressure; Hypertension
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Home BP data will be averaged each month via OmronConnect app on the patients' smartphone, which is programmed to send home BP readings to MyChart via Apple or Google Health.Participants whose home blood pressure reading average is systolic ≥ 130 and diastolic ≥ 80 will trigger the CDS (Clinical Decision Support) tool to assist their physicians with their blood pressure management. Study Team will not be involved in treatment decision making, it will be determined by subject's treating physician. .
  Interventions: Other: Clinical Support Decision Tool
- Usual Care Arm (No Intervention): Physicians will continue to make decisions about the participant's blood hypertension management as usual without the CDS tool.

INTERVENTIONS:
Other: Clinical Support Decision Tool — Participants whose home blood pressure reading average is systolic ≥ 130 and diastolic ≥ 80 will trigger the Clinical Decision Support (CDS) tool to assist their physicians with their blood pressure management. Home BP data will be averaged each month via Omron Connect app on the patients' smartphone, which is programmed to send home BP readings to MyChart via Apple or Google Health. We have designed CDS to present treatment choices of antihypertensive medication regimen based on medications patients are currently taking. For example, patients who are currently taking an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB), our CDS algorithm will recommend addition of a calcium channel blocker as the first tier of recommendation and thiazide diuretics as second tier of recommendation. Laboratory data and home BP in the past month will be presented in a clear and simple manner for the clinicians to activate and use to optimize BP control.
  Arms: Intervention Arm

SUMMARY:
The PCOT study is a multi-site randomized trial of patients 70 years or older with high BP. The main goal of the study Preventing Cognitive Decline by Reducing BP Target Trial (PCOT) is to conduct a large pragmatic clinical trial (PCT) to test the hypothesis that patients who receive care with a combination of clinical decision support (CDS) and team-based care delivered in primary care practices will have better blood pressure control and a lower incidence of mild cognitive impairment and dementia than patients receiving usual medical care. Patients will be recruited from UT Southwestern Medical Center and Parkland Health & Hospital System.

DETAILED DESCRIPTION:
Aim 1 The main aim is to compare the effects of intensive BP intervention between the intervention and usual care arm on the rate of change in TICS-m per year. The investigators will recruit 4,000 patients over 70 years of age with BP >130/80 mmHg from 2 diverse health systems and randomize patients within each health system to usual care or to a combination of care with clinical decision support, practice facilitators and Pharm Ds to lower home BP to < 130/80 mmHg. The primary outcome of this trial will be development cognitive decline as determined by a decrease in TICS-m scores from baseline. As a secondary outcome, the investigators will also measure the development of mild cognitive impairment or dementia in a subset of patients who show a decline of ≥3 points through adjudication.

Aim 2a Determine the potential harms of intensive lowering BP. The investigators aim to recruit 4,000 study participants and compare the effects of lowering home BP below 130/80 mmHg with usual care on hospitalizations, emergency department visits, cardiovascular events, deaths, syncope, falls, fractures, hypotension, electrolyte abnormalities and acute kidney injury. The investigators will capture measures of adherence and health care resource utilization. The investigators will assess QOL in 4,000 patients. The investigators will capture possible harms of lowering BP below 130/80 mmHg. The investigators have chosen clinical outcomes of relevance to all the stakeholders based on prior experience on pragmatic clinical trials and our prior experience in ICD-Pieces. Outcomes will be captured from the telephone assessment by study personnel and electronic health records and/or claims data and reflecting possible harms from all participants will include hospitalizations, emergency department visits, cardiovascular events, deaths, syncope, hypotension, falls, fractures, electrolyte disturbances and acute kidney injury. There will also be capture of adherence by pharmacy refill data. The investigators will capture BP readings from each visit. The investigators will also capture number of encounters with the health system as a measure of health care utilization.

Aim 2b Determine the impact of intensive BP management on QOL. Determine the impact of intensive BP management on QOL. Quality of life (QOL) scores will be obtained using the PROMIS Scale v1.2 - Global Health instrument annually after the administration of the TICS-m.

ELIGIBILITY:
Inclusion Criteria:

* High BP defined as at least 1 BP readings of SBP >= 130 or DBP >=80 during the 24 months prior to enrollment
* Clinic visit with primary care provider within the last 24 months
* Ability to write and speak English or Spanish
* 70 years of age or older
* Ability to understand and willingness to provide informed consent
* Owns a smartphone

Exclusion Criteria:

* Blood pressure consistently <130/80 mmHg
* Presence of dementia, Alzheimer's disease, or significant neurological disease
* Major and unstable heart disease (e.g., acute heart failure (systolic or diastolic), acute on chronic heart failure (systolic or diastolic), acute coronary syndrome or cardiac arrest, liver or renal transplantation
* Under 70 years of age
* Inability to write or speak English or Spanish
* Chronic kidney disease stage 5 or ESKD
* Chemotherapy
* Any conditions judged by the medical providers to contraindicate participation due to risk to patient safety or lack of adherence
* Expected life expectancy under a year

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Decline | 4 years
  Rate of change in Modified Telephone Interview for Cognitive Status (TICS-m) test between study arms. The test has scores ranging from 0 to 42 with higher values indicating better cognitive status.

SECONDARY OUTCOMES:
Mild Cognitive Decline or Dementia | 4 years
  Development of mild cognitive decline or dementia as determined through adjudication from cognitive experts between study arms

OTHER OUTCOMES:
Number of Pharmacy Refills | 4 years
  Between the two groups
Change in quality of life assessment | 4 years
  Quality of life (QOL) scores will be obtained using the PROMIS Scale v1.2 - Global Health instrument annually. The investigators will assess change in quality of life across the four years between the two groups. The Global Health instrument has scores ranging from 4 to 20 for their Mental and Physical Health Items with higher values indiciating better global health.
Number of encounters within the participant's health system | 4 years
  The number of encounters within the participant's respective health system between the two groups will be used to assess healthcare utilization.
Systolic and Diastolic BP Readings | 4 years
  Between the two groups
Combination Pill Use | 4 years
  Between the two groups
BP Above 130/80 | 4 years
  Between the two groups
Count of individuals who experience any of the following safety events: hospitalizations and emergency room visits | 4 years
  Total number of hospitalizations and emergency room visits related to cardiovascular events, syncope, hypotension, falls, fractures, electrolyte disturbances and acute kidney injury between the two groups.
Number of reported deaths | 4 years
  Count of the number of reported deaths between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No